CLINICAL TRIAL: NCT05687240
Title: Effects of QiGong and Tai Chi (QTC) and Heart Rate Variability Biofeedback (HRVB) on Older Adults' Cardiometabolic Risk
Brief Title: Heart Focused Movement Effects on Cardiometabolic Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Linda Larkey, Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00011769
Record Dates: First submitted 2021-06-04; First posted 2023-01-18 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Cardiometabolic Risk Factors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Qigong/Tai Chi Intervention (Active Comparator): Meditative movement practice based on qigong and tai chi, delivered via video link
  Interventions: Behavioral: Qigong/Tai Chi
- Qigong/Tai Chi (QTC) + Heart Rate Variability (HRVB) Intervention (Experimental): Meditative movement practice based on qigong and tai chi, delivered via video link with the addition of a brief practice with a the feedback on heart rate variability from an Inner Balance app.
  Interventions: Behavioral: Qigong/Tai Chi; Behavioral: Heart rate variability biofeedback

INTERVENTIONS:
Behavioral: Qigong/Tai Chi — Participants will engage in 8 weeks of gentle movement/mindfulness videos provided in a daily text prompt, asking that this be practices most days of the week. A choice of practice video links will be provided, ranging from 10-30 minutes in length, and later confirmation texts will be employed to document if practiced, and what length was chosen.
Behavioral: Heart rate variability biofeedback — Randomized participants will be coached to practice a breathing technique that focuses attention on the sensations in the heart area, slowing and deepening the breath, and activating through memory or imagery a positive emotion. This practice is used along with a feedback device that provides information on achievement of the heart rate variability target, "coherence" that represents a neurocardiac state associated with vagal tone, or balance.
  Arms: Qigong/Tai Chi (QTC) + Heart Rate Variability (HRVB) Intervention

SUMMARY:
This study is designed as a two-group parallel randomized controlled trial (N=50) to test effects of 8-weeks of Qigong/Tai Chi (QTC) intervention compared to QTC plus HRVB on HRV parameters (primary), and cardiometabolic risk factors and sequelae (secondary) (e.g., BMI, waist circumference/percent body fat, sleep quality, stress, anxiety/depression, emotional regulation, eating behaviors, and cognitive performance).

DETAILED DESCRIPTION:
Heart rate variability biofeedback (HRVB) will be investigated as a target to optimize Qigong/Tai Chi (QTC) practices based on the expectation that learning to, and practicing changing heart rate variability (HRV) using HRVB, in addition to QTC, will result in higher levels of HRV and coherence than just the QTC alone. This study is designed as a two-group parallel randomized controlled trial to test effects of QTC compared to QTC plus HRVB on HRV parameters (primary), and cardiometabolic risk factors and sequelae (secondary). Fifty participants will be recruited and randomized to one of these groups and receive daily text prompts for 8 weeks to practice (using video links) Tai Chi Easy for 10-30 minutes (length of practice, the participants' choice). Half of the participants randomized to the HRVB enhancement will also be coached to practice HRVB to achieve coherence in their heart beat rhythms prior to practice (QTC plus HRVB group). Data collection at baseline and post intervention will assess body mass index (BMI, waist circumference/percent body fat, sleep quality, stress, eating behaviors, emotion regulation, mood (depression and anxiety), cognitive performance and changes in HRV parameters (high frequency power and coherence).

ELIGIBILITY:
Inclusion Criteria:

* 31.5 inch or above waist circumference women
* 35.5 inch or above waist circumference men
* Has a smartphone or tablet

Exclusion Criteria:

* Those who are unable to stand for 10-minute segments (e.g., wheelchair or walker bound and too weak), and/or unable to walk
* People who have been regularly practicing any form of meditative movement and or HRVB training regularly (i.e., 2 or more times per month for the past 6 months)
* Individuals with diagnosed severe heart arrhythmias, heart transplant, or those with pacemakers would be excluded because either of those interferes with accurately assessing HRV parameters.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Vagal Tone | 8 Weeks
  Measured using resting Heart rate variability and computing parameters of high frequency power and coherence. Will be assessed with participants following a videoguide "to measure their heart rate" that helps them set up equipment and account, seated for 5 minutes of interbeat interval capture using the Inner Balance Bluetooth (HeartMath product) software and earlobe heart beat sensor.

SECONDARY OUTCOMES:
Waist circumference | 8 Weeks
  Waist circumference is measured using tape measure around the waist (after exhale). This is part of the protocol for overall body composition computations using the Marine/Navy protocol.
Abdominal circumference | 8 Weeks
  Abdominal circumference is measured using tape measure around the abdomen/ This is part of the protocol for overall body composition computations using the Marine/Navy Protocol
Height | 8 Weeks
  Measured using tape measure to record inches while participant is standing against a wall.
Weight | 8 weeks
  Digital scales measurement is used to record weight in pounds.
Perceived stress (Perceived Stress Scale-10) | 8 Weeks
  Questionnaire about the amount of stress participants are experiencing daily use includes 10 items with a 0-4 response format. Total scores range from 0-40 with higher scores indicating more perceived stress.
Sleep (Insomnia Severity Index) | 8 Weeks
  Questionnaire about the sleeping habits of participants includes 7 items with response format of 0-4. Total scores range from 0 to 28 with higher scores indicating more severe insomnia: 0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Depression (Profile of Mood States subscale) | 8 Weeks
  Questionnaire includes a 6-item subscale rating level of depression. Participants respond to a single word item by marking a response scale of 0 to 4, with totals ranging from 0-24. Higher scores indicate higher experience of depression.
Anxiety (Profile of Mood States subscale) | 8 Weeks
  Questionnaire includes a 6-item subscale rating level of anxiety. Participants respond to a single word item by marking a response scale of 0 to 4, with totals ranging from 0-24. Higher scores indicate higher experience of Anxiety.
Emotion regulation (Emotion Regulation Questionnaire) | 8 Weeks
  Questionnaire about the emotional regulation of the participants includes 10 items describing ways of regulating emotion with response options from 1-7. Total scores range from 10-70 with higher scores indicating more emotion regulation patterns.
Eating Behaviors (Three Factor Eating Questionnaire) | 8 Weeks
  Questionnaire about the typical eating habits of the participants related to various states of mind or emotions; includes 21 items scored 1-4; total scores range from 21 to 84 with higher scores indicating more controlled/managed and less emotional eating behaviors.
Awareness (one subscale of the Mindful Eating Questionnaire) | 8 Weeks
  The Awareness subscale of the Mindful Eating Questionnaire including 7 items about degree of attention while eating; response format 1-4 (with total score range 7-28) shows higher scores representing more awareness/mindfulness in eating behavior.
Cognitive Performance (Weschler Adult Intelligence Scales -III, letter number sequencing and forward backward digit span tests) | 8 Weeks
  The Letter-number sequencing, and forward backward digit span tests of the Weschler Adult Intelligence Scale (WAIS) III will be administered to study participants to examine cognitive performance. Sets of letters and sets of numbers are read to the participant iteratively; after each set is read, the participant is to repeat back according to instructions to repeat or to repeat in backward order. The first sets are smaller numbers of presented items, increasing with each set of presentations, and are continued until the participant fails a full set. higher scores indicate better cognitive performance. Scores are based on a score of 1 per presented item completed correctly until failure, range 0-51(30 for digits forward/backward and 21 for letter number sequencing).

CONTACTS AND LOCATIONS:
Overall Officials: Linda Larkey, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States